CLINICAL TRIAL: NCT00874458
Title: Ductal Carcinoma in Situ: Protocol Evaluating the Assessment of Extension of Disease by MRI
Brief Title: MRI in Assessing Tumor Size in Women With Ductal Carcinoma In Situ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/25; CALACASS-CCIS; CALACASS-2006/25; 2006-A00251-50 (Other: AFSSAPS ID RCB); INCA-RECF0620
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Experimental)
  Interventions: Procedure: magnetic resonance imaging; Procedure: radiomammography; Procedure: ultrasound imaging

INTERVENTIONS:
Procedure: magnetic resonance imaging
Procedure: radiomammography
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI, may help find ductal carcinoma in situ and find out how far the disease has spread.

PURPOSE: This clinical trial is studying how well MRI works in assessing tumor size in women with ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the contribution of MRI in accurately determining tumor size in women with ductal breast carcinoma in situ (DCIS).

Secondary

* Evaluate the sensitivity of MRI in detecting DCIS.
* Evaluate the contribution of mammography in accurately determining tumor size.
* Compare the contribution of MRI vs mammography in assessing tumor extension.
* Compare the contribution of MRI vs mammography in assessing dense breasts.
* Evaluate the morphology of DCIS by MRI.
* Evaluate the curve of dynamic MRI in assessing DCIS.
* Evaluate the impact of nuclear grade of DCIS by MRI.
* Evaluate the rate of revision surgery.

OUTLINE: Patients undergo clinical examination, mammography, ultrasound imaging, unilateral breast MRI, and tissue sampling.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal breast carcinoma in situ

  * Any grade disease allowed
* Unifocal disease by mammography
* No history of breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WHO performance status 0-2
* Glomerular filtration rate ≥ 30 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No allergy or contraindication to contrast MRI
* No pacemaker or vascular clip

PRIOR CONCURRENT THERAPY:

* No prior or concurrent liver transplantation

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Correlation of tumor extension by MRI with surgical histology | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claire Chapellier, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France